CLINICAL TRIAL: NCT07058272
Title: Effect of PNF Techniques Versus Comprehensive Corrective Exercise Protocol on Pain, Function and Quality of Life in Patients With Upper Cross Syndrome
Brief Title: Effect Of PNF Techniques Versus CCEP On Pain, Function and Quality of Life In Patients With Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-GCUF-079297
Record Dates: First submitted 2025-05-12; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Upper Cross Syndrome
Keywords: Postural Balance; Range of Motion; Muscle Stretching Exercises; Neck Muscles
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Muscle Stretching Exercises; Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization by Chit and Draw Method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): CCEP and TENS
  Interventions: Other: Comprehensive corrective exercise protocol
- Group 2 (Experimental): PNF and TENS
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF) Techniques

INTERVENTIONS:
Other: Comprehensive corrective exercise protocol — Initial phase exercises include lying supine on a foam roll with the arms in 3 different abduction angles, side-lying external rotation, side-lying forward flexion, standing diagonal flexion , and military press .Initial phase lasts for 2 weeks, with exercises progressing from 7 Reps of 10-second holds to 10 Reps of 15-second hold.
  Improvement phase consist of exercises including side-lying external rotation with a dumbbell , side-lying forward flexion with a dumbbell , standing diagonal flexion with a dumbbell, standing external rotation with Thera-Band, standing diagonal flexion with Thera-Band, abduction while sitting on a training ball, prone lying V, T, and W exercises, and standing abduction on a balance board. The improvement phase lasts for 2 weeks, with exercises progressing from seven sets of 10-seconds hold to 10 sets of 15 secs hold.
  The exercises in the maintenance phase are the same as those in the improvement phase, with no increase in intensity and frequency
  Arms: Group 1
Other: Proprioceptive Neuromuscular Facilitation (PNF) Techniques — In this study following PNF Stretching techniques are used
  * Hold-relax or Contract-relax
  * Hold-relax with agonist contraction In the Hold-Relax or Contract-Relax technique, stretching is performed 4sessions per week for each muscle group, with each session lasting 40 min. The protocol includes a 10-sec hold phase followed by a 10-sec contraction phase, repeated for 7 reps . The total duration of this program is 8weeks including 6 weeks of treatment phase and last 2 weeks of detraining.
  In Hold-Relax with Agonist contract, the same procedure is followed as in Hold-Relax method, with 4sessions per week for each muscle group. The patient is asked to hold the initial stretch for 10 sec, followed by a relaxation phase. Afterward, the agonist muscle is contracted to actively move further into the stretch, which is then held for 10 sec. This protocol is performed for 7 reps per session, and the total duration of study is 8 weeks including 6 weeks of treatment program with last 2 weeks
  Arms: Group 2

SUMMARY:
The study aims to determine which approach either PNF Techniques or Comprehensive Corrective Exercise Protocol provides better outcomes for pain relief, functional improvement, and quality of life in patients with upper cross syndrome.

DETAILED DESCRIPTION:
Upper crossed syndrome is caused due to altered muscle activation and movement patterns of the neck, shoulders, head and back muscles. In addition to postural deviations (forward head and rounded shoulders, and an excessive curve of the thoracic spine), upper cross syndrome is characterized by abnormal posture brought on by changed muscle activation patterns and varied movement patterns. Most cases of this condition occurred in people over 20. The symptoms of upper cross syndrome managed by correcting posture, stretching and strengthening the affected muscles, and making ergonomic adjustments.

It will be a Randomized Clinical Trial with sample size of 38. They will be randomly allocated into two groups by using chit and draw method. 19 participants in Group 1 will get PNF protocol while 19 participants in Group 2 get CCEP .For eight weeks, each patient will receive four sessions per week through which their neck disability index, visual analogue scale, and quality of life would measure .Data will be collected at the start of the trial, after four weeks of treatment, and again at the end of treatment. In participants with upper cross syndrome, the goal for applying a comprehensive corrective exercise program and a proprioceptive neuromuscular facilitation technique is to alleviate pain and improve functioning, posture, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age : 25-65
* Symptoms of upper cross syndrome appeared from maximum 6 months
* Occiput to wall test positive
* Patients presenting postural changes e.g: severe kyphosis

Exclusion Criteria:

* Any apparent misalignment in the pelvis or lower limbs.
* Rotation exceeding 5 degrees during forward bending as a result of scoliosis.
* Prior history of joint disorders in the spine, shoulders, and pelvis.
* Body weight that falls outside the normal range (BMI between 18 and 25)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 8 weeks
  NDI comprises 10 items. Each item is rated on a 6-point scale from 0 (no disability) to 5 (complete disability), yielding a total score ranging from 0 to 50. This score can be converted into a percentage by multiplying by 2, resulting in a range from 0% (no disability) to 100% (complete disability).
  Severity Classification:
  0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability 35-50: Complete disability
SF-12 Health Survey | 8 weeks
  The SF-12 Health Survey is a concise, 12-item instrument derived from the SF-36, designed to assess health-related quality of life (HRQoL) across two primary domains: physical health and mental health. It comprises 8 domains. Scores above 50 indicate better health than the average population, while scores below 50 suggest worse health. Each point difference corresponds to a 0.1 standard deviation change

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 8 weeks
  Numerical Pain Rating Scale, used to assess pain intensity. Patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain), providing healthcare providers with a quantifiable measure to evaluate and manage pain.

CONTACTS AND LOCATIONS:
Overall Officials: Usman Iqbal Janjua, Principal Investigator — Ellite College of Managment Sciences, Gujranwala
Locations (1):
- Al-Raee Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (3)Asad, A., Farooq, N., Kafeel, S., Hassan, T., & Zubair, M. (2021). Association of upper crossed syndrome and posture among general population having neck pain in Islamabad. Journal of Rehman Medical Institute, 7(2), 07-11.
- [Background] Seidi F, Bayattork M, Minoonejad H, Andersen LL, Page P. Comprehensive corrective exercise program improves alignment, muscle activation and movement pattern of men with upper crossed syndrome: randomized controlled trial. Sci Rep. 2020 Nov 26;10(1):20688. doi: 10.1038/s41598-020-77571-4. PMID 33244045
- [Background] Chang MC, Choo YJ, Hong K, Boudier-Reveret M, Yang S. Treatment of Upper Crossed Syndrome: A Narrative Systematic Review. Healthcare (Basel). 2023 Aug 17;11(16):2328. doi: 10.3390/healthcare11162328. PMID 37628525